CLINICAL TRIAL: NCT05742542
Title: The Effects of High vs. Low Time Spent Near VO2max During Two Work-matched High Intensity Interval Training.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the State of Santa Catarina (Other)
Responsible Party: Principal Investigator, João Antonio Gesser Raimundo, Member of Human Performance Research Group, University of the State of Santa Catarina
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: VO2maxtrainingUDESantaCatarina
Record Dates: First submitted 2023-02-03; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: VO2max
Keywords: VO2max; Exercise; Aerobic; Performance; Training
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The order of training protocols was randomized and the training programs had a washout period of at least one month.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity interval training with high time spent near VO2max (Experimental): Participants performed high intensity interval training with high time spent near VO2max three times a week for two weeks.
  All training sessions consisted of five times 2 minutes of work and 1 minute of passive recovery. The work intensity was adjusted at 85% and 87% of power output achieved at the end of incremental test for the first and second week, respectively.
  The training sessions were performed using cycle ergometer.
  Findings were compared to high intensity interval training with low time spent near VO2max, which followed the same exercise frequency, intensity and total duration.
  Interventions: Other: Exercise training
- High intensity interval training with low time spent near VO2max (Experimental): Participants performed high intensity interval training with low time spent near VO2max three times a week for two weeks.
  All training sessions consisted of ten times 1 minutes of work and 30 seconds of passive recovery. The work intensity was adjusted at 85% and 87% of power output achieved at the end of incremental test for the first and second week, respectively.
  The training sessions were performed using cycle ergometer.
  Findings were compared to high intensity interval training with high time spent near VO2max, which followed the same exercise frequency, intensity and total duration.
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — Two weeks of high intensity interval training with high or low time spent near VO2max.

SUMMARY:
Maximal oxygen uptake (VO2max) is used to define cardiorespiratory fitness, which is important to health and sport performance in humans. Although different types of training can improve VO2max, the high intensity interval training is recognized as one of the best ways to do it. Furthermore, it has long been speculated that high intensity interval training that elicits a high time spent near VO2max could be the best way to improve VO2max. However, this theory has not been verified. Thus, the investigators performed a randomized controlled trial with crossover in healthy individuals who underwent two high intensity interval training protocols of two weeks, being a workout with longer and other with shorter time spent near VO2max.

DETAILED DESCRIPTION:
Fifteen participants were enrolled in a randomized trial with crossover to perform two weeks of high intensity interval training with high (i.e., five times 2 minutes of work and 1 minute of recovery; T-2min:1min) or low (i.e., ten times 1 minutes of work and 30 seconds of recovery; T-1min:30seg) time spent near VO2max. The work intensity was adjusted at 85% and 87% of power output achieved at the end of incremental test for the first and second week, respectively. Before and after the T-2min:1min and T-1min:30seg, the participants performed tests to determine VO2max, lactate threshold, muscle oxidative capacity, pulmonary oxygen uptake kinetics, power output achieved at the end of incremental test, and power output related to Wingate anaerobic test. The training programs had a washout period of at least one month.

ELIGIBILITY:
Inclusion Criteria:

* Male ≥ 18 years;
* No known musculoskeletal disorders;
* Apparently healthy
* Physically active according to American College of Sports Medicine standards and recommendations (Garber et al., 2011; RIEBE et al., 2015).

Exclusion Criteria:

* Taking any medication that could affect aerobic parameters;
* Smokers;
* Involved in an aerobic training program at the start of the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen uptake | Change at Maximal oxygen uptake after two weeks
  The highest 15 seconds VO2 average determined from rolling averages of 5 seconds samples measured during incremental test or confirmation test of VO2max.

SECONDARY OUTCOMES:
Lactate threshold | Change at Lactate threshold after two weeks
  The work intensity at which blood lactate concentration increased 1 mmol.L-1 above baseline.
Muscle oxidative capacity | Change at Muscle oxidative capacity after two weeks
  Rate recovery of muscle oxygen consumption (k-mV̇O2) of the vastus lateralis, with the k-mV̇O2 indicating muscle oxidative capacity.
Pulmonary oxygen uptake kinetics | Change at Pulmonary oxygen uptake kinetics after two weeks
  The on-transient response for V̇O2 was fitted using a mono-exponential model, which the rate constant (k-pV̇O2) for the kinetics of V̇O2 was calculated as 1/tau (expressed in min-1).
Power output achieved at the end of incremental test | Change at Power output achieved at the end of incremental test after two weeks
  Power output achieved at the end of ramp incremental test (20 W.min-1).
Wingate anaerobic test | Change at Wingate anaerobic test after two weeks
  Peak power, mean power, and minimum power were defined as the highest mechanical power output, the average power sustained throughout the 30-s period, and the power output attained before the end of the test, respectively.
Time spent near VO2max | First to the last day of test or training, an average of 4 weeks
  Time spent at or above 90% or 95% of VO2max.

OTHER OUTCOMES:
Session-rating of perceived exertion | First to the last day of test or training, an average of 4 weeks
  The original 10-point version.
Perceived Recovery Status Scale | First to the last day of test or training, an average of 4 weeks
  The original 10-point version from Laurent et al (2011).
Heart rate | First to the last day of test or training, an average of 4 weeks
  Measured before and during exercise and used to determine 1) the highest heart rate, 2) the time spent near highest heart rate, 3) training impulse, and 4) heart rate variability.
Adipose tissue thickness | Change at Adipose tissue thickness after two weeks
  Adipose tissue thickness measured by a B-mode ultrasound imaging.
Body mass | Change at Body mass after two weeks
  Body mass measured by a digital scale.

CONTACTS AND LOCATIONS:
Overall Officials: João G Raimundo, PhD, Principal Investigator — Member of Human Performance Research Group
Locations (1):
- University of the State of Santa Catarina, Florianópolis, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
The data will be presented as a group (training protocol), but data from representative subjects may be presented if they add relevant information.

REFERENCES:
- [Background] Buchheit M, Laursen PB. High-intensity interval training, solutions to the programming puzzle: Part I: cardiopulmonary emphasis. Sports Med. 2013 May;43(5):313-38. doi: 10.1007/s40279-013-0029-x. PMID 23539308
- [Background] Laursen PB, Jenkins DG. The scientific basis for high-intensity interval training: optimising training programmes and maximising performance in highly trained endurance athletes. Sports Med. 2002;32(1):53-73. doi: 10.2165/00007256-200232010-00003. PMID 11772161
- [Background] Lisboa FD, Raimundo JAG, Salvador AF, Pereira KL, Turnes T, Diefenthaeler F, Oliveira MFM, Caputo F. Acute Cardiopulmonary, Metabolic, and Neuromuscular Responses to Severe-Intensity Intermittent Exercises. J Strength Cond Res. 2019 Feb;33(2):408-416. doi: 10.1519/JSC.0000000000002130. PMID 28704307
- [Background] Lisboa FD, Salvador AF, Raimundo JA, Pereira KL, de Aguiar RA, Caputo F. Decreasing Power Output Increases Aerobic Contribution During Low-Volume Severe-Intensity Intermittent Exercise. J Strength Cond Res. 2015 Sep;29(9):2434-40. doi: 10.1519/JSC.0000000000000914. PMID 26308828
- [Background] Midgley AW, Mc Naughton LR. Time at or near VO2max during continuous and intermittent running. A review with special reference to considerations for the optimisation of training protocols to elicit the longest time at or near VO2max. J Sports Med Phys Fitness. 2006 Mar;46(1):1-14. PMID 16596093
- [Background] Midgley AW, Mc Naughton LR, Wilkinson M. Criteria and other methodological considerations in the evaluation of time at V.O2max. J Sports Med Phys Fitness. 2006 Jun;46(2):183-8. PMID 16823345
- [Background] Raimundo JAG, Turnes T, de Aguiar RA, Lisboa FD, Loch T, Ribeiro G, Caputo F. The Severe Exercise Domain Amplitude: A Comparison Between Endurance Runners and Cyclists. Res Q Exerc Sport. 2019 Mar;90(1):3-13. doi: 10.1080/02701367.2018.1549356. Epub 2019 Jan 17. PMID 30653425
- [Background] Turnes T, de Aguiar RA, Cruz RS, Caputo F. Interval training in the boundaries of severe domain: effects on aerobic parameters. Eur J Appl Physiol. 2016 Jan;116(1):161-9. doi: 10.1007/s00421-015-3263-0. Epub 2015 Sep 15. PMID 26373721